CLINICAL TRIAL: NCT06936670
Title: Effects of High-Resistance Inspiratory Muscle Strength Training on Cardiorenal and Vascular Function in Youth and Young Adults With Type 2 Diabetes
Acronym: IMST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Kalie Tommerdahl, Associate Professor of Pediatrics in the Division of Endocrinology and Diabetes at Seattle Children's Hospital and the University of Washington School of Medicine, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00005096
Record Dates: First submitted 2025-04-14; First posted 2025-04-20 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Type 2 Diabetes; Inspiratory Strength Training; Blood Pressure; Kidney Health; Cardiovascular Function; Diabetic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- IMST (Experimental): Using the POWERBreathe pressure threshold training device, participants will perform 30 inspiratory maneuvers (5 sets of 6, 1 min rest) 6 days/week for 3 months. This is an over the counter product that will be used according to its instructions. The IMST group will train at 75% maximal inspiratory pressure.
  Interventions: Device: Inspiratory Muscle Strength Training (IMST)
- Sham/Placebo (Sham Comparator): Using the POWERBreathe pressure threshold training device, participants will perform 30 inspiratory maneuvers (5 sets of 6, 1 min rest) 6 days/week for 3 months. This is an over the counter product that will be used according to its instructions. The Sham group will train at 15% maximal inspiratory pressure.
  Interventions: Device: Sham Training

INTERVENTIONS:
Device: Inspiratory Muscle Strength Training (IMST) — A novel form of physical training that uses the diaphragm and accessory respiratory muscles to repeatedly inhale against resistance using a handheld device, generating large negative intrathoracic pressures. The device can be set to different levels of resistance, meaning the intervention and sham groups will undergo the same training, but at 75% and 15% of their maximal inspiratory pressure respectively.
  Arms: IMST
Device: Sham Training — The same training regiment but at much lower resistance, offering little to strength training impact.
  Arms: Sham/Placebo

SUMMARY:
High-resistance, short-duration inspiratory muscle strength training (IMST) is a novel lifestyle intervention involving 30 inhalations against a resistive load which requires only ~5 min/day and is thus ideal for youth with T2D (Y-T2D). Investigators seek to 1: assess changes in casual and 24-hr SBP, endothelial function, and arterial stiffness after 3 months of IMST vs. sham training in Y-T2D, 2: Define changes in eGFR andalbuminuria after 3 months of IMST vs. sham in Y-T2D, 3: Interrogate mechanisms of IMST by translational assessments of NO bioavailability, endothelial NO synthase (eNOS) activation, and ROS/oxidative stress, and determine the role of circulating factors.

ELIGIBILITY:
Inclusion Criteria: Aged 14-40, have had T2D for a least one year, HbA1C less than 12%.

-

Exclusion Criteria: Have had type II diabetes for more than 18 years, estimated glomerular filtration rate (eGFR) less than 60 ml/min/1.73m2 or Albumin-to-creatinine ratio (ACR) greater than 2200mg/g, blood pressure greater than 160/100 mm Hg.

-

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 3 months
  Measures of casual clinic and 24-hour ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
Endothelial function | 3 months
  Measured by brachial artery flow-mediated dilation and endothelial cell collection and analysis.
Arterial stiffness | 3 months
  Measured by carotid-femoral pulse-wave velocity and carotid-radial pulse-wave analysis using a SphygmoCor.
Kidney Function | 3 months
  Measured by estimated glomerular filtration rate and albuminuria assessments
Body Composition | 3 months
  Measured by BIS (Bioimpedance spectroscopy)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medicine Diabetes Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided